CLINICAL TRIAL: NCT02680405
Title: Identification of Epidermal Signatures in Patients With Atopic Dermatitis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Jewish Health (Other)
Collaborators: MedImmune LLC (Industry)
Responsible Party: Principal Investigator, Donald Leung, MD, PhD, MD, PhD, National Jewish Health
Other Study IDs: HS-2930
Record Dates: First submitted 2016-01-29; First posted 2016-02-11 (Estimated); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Skin biopsy, blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Atopic Dermatitis: Subjects with Atopic Dermatitis will have blood draw, skin biopsies and tape stripping
  Interventions: Procedure: Skin Biopsy; Procedure: Skin tape stripping; Procedure: Blood draw
- Non Atopic Dermatitis: Subjects with no Atopic Dermatitis will have blood draw, skin biopsies and tape stripping
  Interventions: Procedure: Skin Biopsy; Procedure: Skin tape stripping; Procedure: Blood draw

INTERVENTIONS:
Procedure: Skin Biopsy — Full thickness skin biopsies will be collected from each subject used for proteomic and genomic analysis of associated biomarker levels.
Procedure: Skin tape stripping — Skin tape stripping used for proteomic and genomic analysis of associated biomarker levels.
Procedure: Blood draw — Whole blood and serum testing used for proteomic and genomic analysis of associated biomarker levels.

SUMMARY:
Atopic dermatitis is a skin disorder with an itchy, red skin rash. This may be because certain proteins are increased in the skin of AD patients. The increased expression of these proteins play an important role in the development of AD and may increase the risk for persons with AD to get skin infections and allergies.

There are very few non-invasive ways to diagnose and monitor the development and progression of atopic dermatitis. The goal of this study is to develop laboratory tests, done on skin samples collected by tapy stripping, that can be used for early detection and monitoring the response to treatment for a variety of skin diseases, including atopic dermatitis.

DETAILED DESCRIPTION:
Atopic dermatitis (AD) is a highly pruritic, chronic inflammatory skin disease that affects up to 25% of children and 10% of adults. Atopic skin disease is associated with significant morbidity as well as physical, psychological, and economical quality-of-life impairment. The economical impact of AD and the requirement for family support can be extraordinary and may be greater than what is typically found for asthma and type I diabetes, respectively. In many patients, the early onset of AD is the first clinical manifestation of allergic disease and often triggers the atopic march, the subsequent development of food allergy, allergic rhinitis, and asthma. The skin of AD patients is characterized by an increased Th2 axis, cellular infiltration and significant epithelial inflammation. These factors permit increased penetration of invading allergens and pathogens that further drive AD pathogenesis and pruritus (itch). Approximately 90% of AD patients are colonized with S. aureus, while only 5 - 30% of non-atopic individuals are colonized. Novel therapeutic approaches are currently in clinical trials which provide the opportunity to target pathways integral to AD disease pathogenesis. In recent years, it has been shown that AD is more heterogeneous than initially perceived. Since novel therapeutics target different pathways, one therapeutic approach may not work for all AD patients and each therapy may provide a different level of clinical benefit. Additionally, since AD manifests primarily in the skin, blood collection and analysis may not be the most indicative measurement to determine which therapy is best for each patient. Despite improved understanding of AD, validated methods to non-invasively diagnose and monitor the development or progression of AD are sorely lacking. Additionally, a non-invasive method is needed to understand inflammation at the site of disease manifestation and potentially identify which biological pathways are most relevant for a given patient. This will allow a more personalized approach to treatment of patients with AD.

The investigator has hypothesized that skin proteins are differentially expressed in the upper layers of disease versus non-disease skin tissue and that these may be used as biomarkers for skin changes linked to the development of AD. Previously a method for comparing expression of skin proteins by extracting proteins from tape strips and evaluating differences using mass spectrometry-based proteomics was developed. This non-invasive method is suitable for use in all AD patients and has been used to show an increase in specific skin proteins in AD patients versus normal controls. Despite this success, additional studies are needed to compare gene and protein expression obtained from tape strips with genomic and proteomic profiles from full thickness skin and whole blood. This proposed study will determine the validity of using non-invasive tape stripping, as a surrogate for skin biopsy and whole blood collection, to identify the inflammatory pathway most up-regulated in a given AD patient. This information will be used in defining biomarkers that will facilitate personalized medicine approaches using emerging novel therapeutics.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained prior to any study related procedure taking place.
2. Male or Female age 18-65 years inclusive at the time of screening
3. Current disease state meeting the Hanifin and Rajka criteria for AD Or Non-atopic with no history of skin disease
4. Atopic dermatitis that affects ≥ 15% body surface area (BSA)
5. No clinically significant abnormality on the basis of medical/medication history or physical examination

Exclusion Criteria:

Subjects who meet any of the following criteria will not be eligible:

1. Active dermatologic conditions which may confound the diagnosis of AD or would interfere with assessment of treatment, such as scabies, seborrheic dermatitis, cutaneous lymphoma, ichthyosis or psoriasis
2. Known active allergic or irritant contact dermatitis
3. Use of topical corticosteroids or humectants (e.g. containing urea or lactic acid) within 7 days of Visit 1 and throughout the study. Standard occlusives and emollients are permitted
4. Treatment of AD with a medical device (e.g. Atopiclair®, MimyX®, Epicerum®, Cerave®, etc) within 7 days of Visit 1 and throughout the study. Standard occlusive and emollients are permitted.
5. Use of tanning beds or phototherapy within 8 weeks
6. Receipt of any marketed or investigational biologic agent within 4 months or 5 half-lives prior to Visit, whichever is longer
7. Receipt of any investigational non-biologic agent within 3 months or 5 half-lives prior to Visit, whichever is longer
8. Treatment with the following medications within the last 4 weeks prior to Visit:

   * systemic immunosuppressive/immunomodulating drugs ((eg, methotrexate, cyclosporine, azathioprine, mycophenolate mofetil, tacrolimus, interferon gamma, intramuscular long-acting depot corticosteroid).)
   * Systemic corticosteroid use (excludes topical, inhaled, or intranasal delivery)
   * Topical calcineurin inhibitor use
9. Known history of allergy or reaction to tape or adhesives
10. Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will enroll up to 50 participants who are 18 to 65 years of age. Up to 40 of the participants will have Atopic Dermatitis. Up to 10 of the participants will not have Atopic Dermatitis. Approximately 25 of the participants will be women and 25 will be men.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-04; Primary Completion 2016-07 (Actual); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Epidermal Barrier Expression Levels | 2.5 years
  * Expression level of filaggrin in the epidermis
  * Expression level of TSLP in the epidermis
  * Expression level of Corneodesmosin in the epidermis
  * Expression level of Serpin B3 in the epidermis

CONTACTS AND LOCATIONS:
Overall Officials: Donald Leung, MD, PhD, Principal Investigator — National Jewish Health
Locations (1):
- National Jewish Health and University of Colorado Denver, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
The investigator will not provide results of any tests performed for this study to the participant.